CLINICAL TRIAL: NCT01104363
Title: Prosthetic Fit Improving With Splint Implant Impressions: Double-blind, Randomised Clinical Trial of Accuracy and Materials.
Brief Title: Splint Versus Non-splint Implant Impressions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical commentate has not be obtained by the institution.
Sponsor: Hospital San Pietro Fatebenefratelli (Other)
Collaborators: Nobel Biocare (Industry)
Responsible Party: Principal Investigator, Marco Tallarico, Principal investigator, Hospital San Pietro Fatebenefratelli
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NobelBiocare-RCT-Procera
Record Dates: First submitted 2010-04-02; First posted 2010-04-15 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Dental Implants; Dental Impression Materials; Dental Impression Techniques
Keywords: Dental implants
MeSH Terms: interventions — poliovirus receptor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Snow white Plaster 2 (Experimental): Test
  Interventions: Procedure: Snow white plaster 2
- Primopattern LC gel + PVS (Active Comparator): Control
  Interventions: Procedure: Primopattern LC gel + PVS

INTERVENTIONS:
Procedure: Snow white plaster 2 — Test. Plaster impression not splinted.
  Arms: Snow white Plaster 2
Procedure: Primopattern LC gel + PVS — Control PVS impression
  Arms: Primopattern LC gel + PVS

SUMMARY:
The purpose of this study is to evaluate the effectiveness of heavy Vinyl PolySiloxane (VPS) and splinted implants impression (Study Group, SG) technique versus plaster implant impression (Control Group, CG) technique, in 12 edentulous patients rehabilitated with the All-on-4/6 concept and Procera® Implant Bridge (P.I.B.). A longitudinal, double blinded, randomised clinical trial (RCT) was designed to evaluate the accuracy of the impression. All patients were monitored from implant placement until prosthetic loading.

DETAILED DESCRIPTION:
The aim of the present study was to investigate the accuracy of pick-up, splinted implants, and heavy VPS impression techniques (Aquasil Putty DECA™ and Aquasil Ultra Light Viscosity (LV) Regular Set, Dentsply International Inc, Caulk, USA); to compare two splint materials for implants: Primopattern LC gel (Primotec, Bad Homburg, Germany), and Smart Dentin Replacement (SDR™, Dentsply International Inc, Caulk, USA); to examine the clinical factors affecting the accuracy of implant impressions; to test the tension-free fit of the new scanner and software NobelProcera™ (NobelBiocare, AB, Göteborg, Sweden) titanium frameworks.The hypothesis to demonstrate is that all impression techniques and used materials reduce time for final restoration and improve the accuracy of the impression.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older.
* Both genders.
* Fully edentulous patients.
* Both maxilla and mandible.
* Dental implant rehabilitation utilizing the All-on-4 concept at least 8 weeks before impression.
* External hex dental implant.
* Patients with ability to understand and sign the informed consent prior to starting the study.
* Adequate oral hygiene.
* Immediate functional loading.
* Implant stability quote value =/> 65 from implant placement to final prosthetic rehabilitation.

Exclusion Criteria:

* Failure of one or more inclusion criteria.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Implant failure | Up to 5 years after implant placement
  An implant was consid- ered to be a failure if it was lost owing to mobility, implant fracture and/or any infection requiring implant removal.

SECONDARY OUTCOMES:
Inter-implants distance between groups | 4 to 5 months after implant placement (baseline)
  Inter-implants distance between groups assessed both on casts and digital photos measured in mm.
Chair-time | 4 to 5 months after implant placement (baseline)
  Time needed to take impression in both control and test group measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tallarico, dr., Study Director — Private Practice
Locations (2):
- Italy (2):
  - Marco Tallarico, Rome, RM
  - Studio odntoiatrico specialistico dr. Marco Tallarico, Rome, RM

REFERENCES:
- [Background] Lee H, So JS, Hochstedler JL, Ercoli C. The accuracy of implant impressions: a systematic review. J Prosthet Dent. 2008 Oct;100(4):285-91. doi: 10.1016/S0022-3913(08)60208-5. PMID 18922257